CLINICAL TRIAL: NCT03012555
Title: Nutritional Vitamin D3 in Patients With Sickle Cell Disease
Brief Title: Vitamin D3 in Patients With Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 13-1056
Record Dates: First submitted 2017-01-04; First posted 2017-01-06 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Vitamin D
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Sickle Cell Disease and Vitamin D deficiency

SUMMARY:
There are approximately 90,000 individuals in the United States with sickle cell disease (SCD). Studies have shown that up to 98 percent of patients with Sickle Cell Disease have a vitamin D deficiency, defined as a 25-hydroxyvitamin D level (25(OH)D) less than or equal to 20 ng/mL. As a result, of low bone density, patients may develop osteonecrosis, chronic inflammation and related pain. This study will be coordinated with patients' regularly scheduled visits for medical care and will require patients to submit blood sample at the start of the study and at 3, 6, 9, AND 12 month visits. Patients will also be scheduled for a bone density measurement (DXA scan) at the start of the study and after 12 months of supplementation to assess for any bone re-mineralization. Thus, the main purpose of this study is to find the amount of nutritional vitamin D that needs to be taken by patients with sickle cell disease in order to correct vitamin D deficiency. The study will also test whether vitamin D supplements improve bone health and reduce inflammation.

DETAILED DESCRIPTION:
This is an observational cohort study to follow vitamin D levels over time in patients with sickle cell disease receiving doses of vitamin D as part of their clinical care for vitamin D deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years and older)
* Diagnosis of sickle cell disease by hemoglobin electrophoresis (HbSS, hematopoietic blood stem cell [HbSC], Sickle cell b0 Thalassemia, Sickle cell b+ Thalassemia)
* Able to give informed consent
* Any race/ethnicity/socioeconomic status

Exclusion Criteria:

* Pediatric patient (less than 18 years of age)
* Unable to give informed consent
* Untreated primary hyperparathyroidism (ICD9 codes 252.01XX and 252.00XX)
* hypercalcemia (serum calcium level > 11 mg/dl; ICD9 codes 275.42XX, 259.3XX, 252.00F)
* Pregnancy: a urine pregnancy test, or a serum pregnancy test, will be obtained at the time of enrollment in addition to reviewing the medical record; pregnant patients will be excluded because they should not undergo DXA scanning
* Patients taking atorvastatin, thiazide diuretics and digoxin, which are medications that can interact with vitamin D
* Non-English speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult Patients (18 years and older) with a diagnosis of sickle cell disease by hemoglobin electrophoresis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-10; Primary Completion 2016-08-11 (Actual); Study Completion 2016-08-11 (Actual)

PRIMARY OUTCOMES:
25(OH)D level | 12 months
  Amount of vitamin D to correct vitamin D deficiency in patients with sickle cell disease

SECONDARY OUTCOMES:
Dexa Scan | 12-18 months
  Change in bone remineralization after 12 months of vitamin D supplementation
CRP level | 12 months
  Medical record abstraction for CRP levels to indicate changes in inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Jena Simon, MS, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States